CLINICAL TRIAL: NCT04145167
Title: Prospective Evaluation of Treatment Strategies in Patients Presenting With Chronic Total Occlusions at Coronary Angiogram
Brief Title: Observational Registry on Clinical Outcome After Diagnosis of Chronic Total Occlusions
Acronym: PETS-CTO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziekenhuis Netwerk Antwerpen (ZNA) (Other)
Responsible Party: Principal Investigator, Pierfrancesco Agostoni, Dr, Ziekenhuis Netwerk Antwerpen (ZNA)
Other Study IDs: EC 5269
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Chronic Total Occlusion of Coronary Artery; Angina Pectoris
Keywords: chronic total occlusion; coronary percutaneous intervention; ischemic heart disease
MeSH Terms: conditions — Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Medical Treatment: This group will include all patients with a diagnose of coronary chronic total occlusions who will be treated by medical therapy only, for any clinical/angiographic/instrumental indication.
- Percutaneous intervention: This group will include all patients with a diagnose of coronary chronic total occlusions who will be treated by percutaneous intervention (CTO-PCI), as indicated by the heart-team.
- Surgical treatment: This group will include all patients with a diagnose of coronary chronic total occlusions (generally not isolated) who will be treated by means of coronary artery by-pass grafting (CABG), as indicated by heart-team decision.

SUMMARY:
This registry aims at enrolling all consecutive patients presenting with at least one chronic total occlusion at coronary angiogram as diagnosed during angiography in our catheterization laboratory during 1 year.

All patients will undergo - whenever possible - a cardiopulmonary excercise test and a non-invasive investigation for myocardial ischemia/viability (by means of echo-dobutamine stress test or perfusion scintigraphy or cardiac magnetic resonance) prior to any eventual revascularization therapy. All patients - including those treated by medical therapy only - will repeat the same investigations after one year of follow-up. In addition to these investigations, clinical outcome and quality of life (including the Seattle Angina Questionnarie and a dedicated depression questionnaire) will be evaluated at baseline and at follow-up.

Primary objective of this study is to investigate the improvement in physical conditions (as expressed by the performance at follow-up CP test), the reduction in ischemia (as evaluated by follow-up non-invasive imaging tests) and the severity of angina according to clinical assessment (including Seattle Angina Questionnaires [SAQ], Canadian Class Score[CCS] and 6-mins walking test).

DETAILED DESCRIPTION:
Background The clinical benefits of performing chronic total occlusion (CTO) percutaneous coronary intervention (PCI) represent still a matter of debate in the community of interventional cardiologists[1]. Improvements in terms of symptoms' relief after successful CTO recanalization are growing, with emerging data from randomized clinical trials (RCT) [2] in addition to the already existing large registries[3,4]. In addition, these registries offer data supporting reduction in hard clinical endpoints - including incidence of myocardial infarction (MI) and cardiac death - which however, has so far not been confirmed in RCT. Furthermore, data regarding reduction in ischemia burden after successful CTO-PCI - despite intuitive - and its clinical implications are still lacking, with only a small registry[5] reporting on improved Cardiopulmonary Exercise parameters after successful CTO recanalization. It's also widely known that chronic (refractory) angina significantly impacts the daily life of patients with CTO lesions, not only affecting their quality of life, but also leading to a de-conditioning and a self-limitation in daily activities, creating a negative loop that further reduce the efforts tolerance in these delicate patients. Moreover, recent data suggest that incidence of depression is common among patients with known coronary CTO, and that benefits from successful CTO-PCI may include improvements in psychological health[6].

Of note, the outcome of patients presenting with CTO lesions has been so far investigated only in selected groups of populations (including those with evidence of ischemia/viability, those undergoing CTO-PCI procedures…). However, a systematic and prospective analysis of all consecutive patients presenting with CTO lesions during coronary angiogram, independently by any therapeutic strategy, is so far lacking.

Objective Aim of this registry is to include all consecutive patients presenting with CTO lesion in a relevant coronary vessel (or relevant side branch [namely any coronary vessel with diameter ≥2.5mm]) during cardiac catheterization, to comprehensively analyse their characteristics and to investigate the clinical outcome at 1 year, independently of their therapeutic work-up.

Methodology All patients undergoing coronary angiogram in our centre will be screened for eligibility in the registry. Inclusion and exclusion criteria are here reported.

Inclusion Criteria:

* Presence of at least one untreated CTO at basal angiography (defined as a total occlusion in any major coronary vessel or relevant side branches [reference vessel diameter ≥2.5mm or as judged by two independent interventional cardiologists], with TIMI 0 in the distal segment and at least 3 months old - according to clinical information or of unknown age).
* In patients with history of CABG, a CTO can be included when the occlusion is located in a vessel without a graft in the distal vessel or in case of graft occlusion.
* Age > 18 years
* Willing to participate and able to understand, read and sign the informed consent document after the diagnostic procedure

By study design, no specific exclusion criteria are indicated, except for the lack of will to participate in the study or inability to provide informed consent (e.g. by patient admitted with cardia arrest or unconscious).

Written informed consent form will be collected in all patients.

Withdrawal criteria Patients will be able to withdraw from the study at any time at their request.

Briefly, all patients fulfilling the inclusion criteria will be enrolled in this registry. Of note, the relevance of the CTO-vessel will be adjudicated by two different experienced interventional cardiologists. CTO of small vessels without haemodynamic relevance will not be included in this study. After evaluation in a dedicated CTO-outpatient clinic, they will undergo a cardiopulmonary exercise test (Baseline CP test) and MIBI-scan before any therapeutic strategy (including CTO-PCI or surgical revascularization).

After one year from the enrolment, patients will be evaluated again in the dedicated outpatient clinic, with repeated imaging and functional tests.

Study Objective Primary objective of this study is the improvement in physical conditions as expressed by the performance at follow-up CP test, the reduction in ischemia as evaluated by follow-up MIBI-scan and the severity of angina according to clinical assessment (including Seattle Angina Questionnaires [SAQ], Canadian Class Score[CCS] and 6-mins walking test). Quality of life will also be assessed by means of a dedicated Depression score. These outcomes will be stratified according to the therapeutic strategy adopted in each patient (namely optimal medical treatment alone, CTO-PCI or surgical revascularization).

Secondary endpoints will include a composite of major adverse clinical events (defined as cardiovascular death, myocardial infarction and ischemia-driven revascularization), re-hospitalization for angina/heart-failure, bleeding episodes, strokes and need for specialist/non-specialist outpatient evaluation because angina in the study period.

Sample Sizing By study design, all consecutive patients presenting with relevant CTO lesions at coronary angiogram will be included in the analysis. Given the explorative nature of this registry (at present no similar studies are available in the literature), a solid sample-sizing cannot be performed.

Considering the reported incidence of CTO lesions - ranging from 15-25% of the coronary angiographies performed - and the procedure-volume of this centre (approximately 4000 coronary angiograms per year), a 1-year of consecutive enrolment should provide a large number of subjects (approximately 600) to investigate with solidity eventual significant improvements in the primary endpoints.

Previous registries have reported on the outcome of CTO-PCI procedures in terms of CPET parameters, enrolling approximately 30 patients [7], however given the purely observational nature of this study and the fact the many patients could result not eligible to perform an exercise test (similarly for the echo-stress investigation), a large patient pool has been selected for the present registry, in order to provide solid data for this analysis and a possibly clear response to this unresolved clinical controversy.

Duration of the study (per patient) The duration of participation for each patient will be approximately 1 year. Patients presenting with evidence of CTO lesions at angiography will be screened and, if meeting the study eligibility criteria, will be enrolled in the study. A comprehensive clinical evaluation, together with cardiopulmonary exercise test and MIBI-scan will be performed in the month following the enrollment. Independently of the subsequent treatment strategies, patients will be followed-up for 1 year, including a new clinical evaluation in outpatient setting with cardiopulmonary test and MIBI-scan at the end of the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one untreated CTO at basal angiography (defined as a total occlusion in any major coronary vessel or relevant side branches [reference vessel diameter ≥2.5mm or as judged by two independent interventional cardiologists], with TIMI 0 in the distal segment and at least 3 months old - according to clinical information or of unknown age).
* In patients with history of CABG, a CTO can be included when the occlusion is located in a vessel without a graft in the distal vessel or in case of graft occlusion.
* Age > 18 years
* Willing to participate and able to understand, read and sign the informed consent document after the diagnostic procedure

Exclusion Criteria:

* Lack of will to participate in the study or inability to provide informed consent (e.g. by patient admitted with cardiac arrest or unconscious)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes all patients aged >18 with coronary artery disease undergoing coronary catheterization. Key condition to be enrolled in the registry is the evidence of chronic total occlusion and the will to participate in the study.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in ischemia and angina paramteres | 1 year
  Parameters of Cardiopulmonary Exercise test, non-invasive imaging tests and angina questionnaires.

SECONDARY OUTCOMES:
Composite of major adverse clinical events | 1 year
  Composite of cardiac death, myocardial infarction and ischemia-driven revascularization.
Re-hospitalization | 1 year
  Episodes of re-hospitalization due to angina/heart-failure
Outpatient clinic evaluation | 1 year
  Need for specialist/non-specialist outpatient evaluation because angina

CONTACTS AND LOCATIONS:
Locations (1):
- ZNA Middelheim, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tajti P, Brilakis ES. Chronic Total Occlusion Percutaneous Coronary Intervention: Evidence and Controversies. J Am Heart Assoc. 2018 Jan 12;7(2):e006732. doi: 10.1161/JAHA.117.006732. No abstract available. PMID 29330258
- [Background] Werner GS, Martin-Yuste V, Hildick-Smith D, Boudou N, Sianos G, Gelev V, Rumoroso JR, Erglis A, Christiansen EH, Escaned J, di Mario C, Hovasse T, Teruel L, Bufe A, Lauer B, Bogaerts K, Goicolea J, Spratt JC, Gershlick AH, Galassi AR, Louvard Y; EUROCTO trial investigators. A randomized multicentre trial to compare revascularization with optimal medical therapy for the treatment of chronic total coronary occlusions. Eur Heart J. 2018 Jul 7;39(26):2484-2493. doi: 10.1093/eurheartj/ehy220. PMID 29722796
- [Background] Tomasello SD, Boukhris M, Giubilato S, Marza F, Garbo R, Contegiacomo G, Marzocchi A, Niccoli G, Gagnor A, Varbella F, Desideri A, Rubartelli P, Cioppa A, Baralis G, Galassi AR. Management strategies in patients affected by chronic total occlusions: results from the Italian Registry of Chronic Total Occlusions. Eur Heart J. 2015 Dec 1;36(45):3189-98. doi: 10.1093/eurheartj/ehv450. Epub 2015 Sep 2. PMID 26333367
- [Background] Jang WJ, Yang JH, Choi SH, Song YB, Hahn JY, Choi JH, Kim WS, Lee YT, Gwon HC. Long-term survival benefit of revascularization compared with medical therapy in patients with coronary chronic total occlusion and well-developed collateral circulation. JACC Cardiovasc Interv. 2015 Feb;8(2):271-279. doi: 10.1016/j.jcin.2014.10.010. PMID 25700750
- [Background] Abdullah SM, Hastings JL, Amsavelu S, Garcia-Morales F, Hendrix F, Karatasakis A, Danek BA, Karacsonyi J, Rangan BV, Roesle M, Khalili H, Banerjee S, Brilakis ES. Percutaneous Coronary Intervention of Coronary Chronic Total Occlusions Improves Peak Oxygen Uptake During Cardiopulmonary Exercise Testing. J Invasive Cardiol. 2017 Mar;29(3):83-91. PMID 28255103
- [Background] Yeh RW, Tamez H, Secemsky EA, Grantham JA, Sapontis J, Spertus JA, Cohen DJ, Nicholson WJ, Gosch K, Jones PG, Valsdottir LR, Bruckel J, Lombardi WL, Jaffer FA. Depression and Angina Among Patients Undergoing Chronic Total Occlusion Percutaneous Coronary Intervention: The OPEN-CTO Registry. JACC Cardiovasc Interv. 2019 Apr 8;12(7):651-658. doi: 10.1016/j.jcin.2018.12.029. Epub 2019 Mar 13. PMID 30878475
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Derived] Poletti E, Zivelonghi C, Castaldi G, Vermeersch P, Convens C, Selleslagh P, Prihadi E, Droogmans S, Scott B, Agostoni P. Prospective Evaluation of Treatment Strategies in Patients Presenting With Chronic Total Occlusion: The PETS-CTO Registry. Catheter Cardiovasc Interv. 2025 Jul;106(1):443-453. doi: 10.1002/ccd.31559. Epub 2025 Apr 28. PMID 40296468